CLINICAL TRIAL: NCT06465810
Title: A Non-interventional, Prospective, Multi-country Study Collecting Real-world Data on the Characteristics, Treatment Patterns, and Outcomes of Patients With Transthyretin (ATTR) Amyloidosis
Brief Title: Non-interventional Study of Patients With Transthyretin (ATTR) Amyloidosis
Acronym: MaesTTRo
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: D8450R00003
Record Dates: First submitted 2024-05-13; First posted 2024-06-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Transthyretin Amyloidosis; ATTR-CM; ATTRv-PN; ATTR; ATTR-Mixed; hATTR
Keywords: Amyloidosis; Transthyretin; Hereditary transthyretin-mediated (hATTR) amyloidosis; hATTR amyloidosis; Hereditary ATTR amyloidosis; Wild-type amyloidosis; wtATTR amyloidosis; ATTRv amyloidosis; ATTRwt amyloidosis; Polyneuropathy; Familial amyloid polyneuropathies; ATTR; Transthyretin amyloidosis; TTR-mediated amyloidosis; Polyneuropathies; Amyloid neuropathies; Amyloid neuropathies, familial; Amyloidosis, familial; Eplontersen; Non-interventional; Observational; Real-world
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis; Amyloid Neuropathies, Familial; Polyneuropathies; Amyloid Neuropathies; Amyloidosis, Familial | interventions — Amyloid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ATTR cardiomyopathy (ATTR-CM): Patients with ATTR-CM at enrollment
  Interventions: Drug: Treatment of transthyretin (ATTR) amyloidosis in observational study setting
- Hereditary polyneuropathy (ATTRv-PN): Patients with ATTRv-PN at enrollment
  Interventions: Drug: Treatment of transthyretin (ATTR) amyloidosis in observational study setting
- ATTR-Mixed: Patients with a mixed ATTR amyloidosis phenotype
  Interventions: Drug: Treatment of transthyretin (ATTR) amyloidosis in observational study setting

INTERVENTIONS:
Drug: Treatment of transthyretin (ATTR) amyloidosis in observational study setting — Data will be collected on patients with ATTR amyloidosis in a real-world setting

SUMMARY:
The MaesTTRo study aims to enroll a global cohort of patients with transthyretin (ATTR) amyloidosis to longitudinally observe the natural course of the disease and describe real-world treatment patterns and outcomes. In addition, information on the effectiveness of ATTR amyloidosis treatments, including eplontersen, which is a ligand-conjugated antisense oligonucleotide gene silencing treatment targeting activity against both the mutant and wild-type TTR protein, will be collected.

DETAILED DESCRIPTION:
MaesTTRo is an international, longitudinal, non-interventional study of adult patients with transthyretin (ATTR) amyloidosis.

The study plans to enroll a minimum of 1850 patients with ATTR amyloidosis, including a minimum of 850 patients with ATTR cardiomyopathy (ATTR-CM), and a minimum of 100 patients with ATTRv-PN hereditary polyneuropathy.

The enrollment period is expected to last approximately 4 years. The duration of follow-up for each patient will be at least 3 years and up to 7 years depending on the date when the patient is enrolled.

This study design will include both primary and secondary data. Primary data will consist of patient-reported outcome (PRO) questionnaires. Patients will be asked to complete electronic PRO questionnaires at enrollment and every 6 months (±3 months) only during routine visits. Secondary data will consist of demographic, clinical, and treatment information, and will be collected as per routine clinical practice. These data will be abstracted directly from the electronic health record or review of paper charts for each patient and entered in the electronic data capture system. No site visits are required for this study, and patients will not be contacted for data collection outside of routine clinic visits.

For patients enrolled in the United States, a tokenization process (creation of a unique, encrypted identifier called a token, in place of personal identifiable information) will be used to collect additional de-identified data (e.g., healthcare resource use, healthcare costs) from other sources that are part of patients' routine medical care (electronic medical, hospital, or pharmacy records). Only de-identified data will be analyzed. Patients will be given a choice within the informed consent form to opt in or opt out of participating in the tokenization process.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to provide written informed consent to participate in the study
* Confirmed diagnosis of amyloid transthyretin (ATTR) amyloidosis
* Aged ≥18 years at the time of signing the informed consent
* Patient willing and able to participate in collection of electronic patient reported outcomes (PROs)

Exclusion Criteria:

* Concurrent participation in any interventional trial for ATTR amyloidosis
* Involvement in the planning and/or conduct of the current study
* Patients with evidence of primary or light chain amyloidosis (AL) or serum protein A amyloidosis (AA)
* Asymptomatic patients with ATTR amyloidosis and asymptomatic ATTR mutation carriers

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of amyloid transthyretin (ATTR) amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2031-12-29 (Estimated); Study Completion 2031-12-29 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  * Age
  * Sex as determined by the investigator (male/female)
  * Race and ethnicity, where allowed
Treatment patterns (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following treatments will be assessed:
  * ATTR amyloidosis treatment: Tafamidis, Diflunisal, Acoramidis, Vutrisiran, Patisiran, Inotersen, Eplontersen, Doxycycline and taurodesoxycholic acid, Liver transplant
  * Heart failure/arrhythmia-related treatment: Diuretics, Angiotensin converting enzyme inhibitor, Angiotensin receptor blocker, Angiotensin receptor-neprilysin inhibitor, Anticoagulation, Beta-blockers, Sodium-glucose co-transporter-2 inhibitor, Mineralocorticoid receptor antagonist, Digoxin, Pacemaker use, Implantable cardioverter-defibrillator, Left ventricular assist device, Cardiac transplant, Transcatheter aortic valve replacement, Surgical aortic valve replacement
  * Polyneuropathy-related treatment: Antiepileptics (gabapentin, pregabalin, carbamazepine, phenytoin), Antidepressants, Topical pain treatments, Opioids, Tetrahydrocannabinol
  * Other: Medications for gastrointestinal symptoms, Vitamin A supplementation, Dialysis
Clinical characteristics (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following clinical characteristics will be assessed:
  * Modified body mass index (mBMI)
  * Medical history
  * TTR genetic test results
  * Family history of ATTR
  * Time period between the first symptoms to date of diagnosis of ATTR
  * Time since diagnosis of ATTR
Findings from biopsy (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following biopsy information will be collected:
  * Type of biopsy
  * Amyloid identification result (Positive, Negative, Inconclusive for amyloid)
  * Method of amyloid typing
  * Result of the biopsy (Normal/Abnormal)
  * Reason for considering the biopsy result abnormal
Findings from Cardiovascular magnetic resonance imaging (CMR) (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following information will be collected: extracellular volume (ECV), contrast use, left ventricular (LV) end-diastolic volume, LV end-systolic volume, LV ejection fraction, LV Mass Index, interventricular wall thickness, right ventricular Free Wall Thickness, LV Free Wall Thickness, left Atrial Volume Index, native T1 mapping, CMR result (Normal/Abnormal), reason for considering the result abnormal.
Findings from Bone tracer cardiac scintigraphy (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following information will be collected: Type of tracer, Heart to contralateral lung ratio (H/CL), Perugini grade, scintigraphy result (Normal/Abnormal), reason for considering the result abnormal.
Findings from Echocardiography (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following information will be collected: LV ejection fraction, LV End Diastolic Volume, LV End Systolic Volume LV End Diastolic Dimension, LV End Systolic Dimension, Interventricular Septal Thickness End Diastole, Posterial Wall Thickness End Diastole, Left Ventricular Mass Index, Left Atrial Volume, Left Atrial Volume Index, Mitral valve regurgitation, Aortic valve regurgitation, Tricuspid valve regurgitation, Pulmonic valve regurgitation, LV Outflow Gradient, Stroke Volume, Lateral early diastolic myocardial velocity (e' lateral), Medial early diastolic myocardial velocity (e' medial), Mitral E/e' Ratio, Early diastolic mitral inflow velocity (E), Late diastolic mitral inflow velocity (A), Mitral Peak E/A Ratio, Global LV longitudinal strain, Pulmonary artery systolic pressure, RV Free Wall Thickness Severity of Aortic stenosis, Severity of Mitral stenosis.
ECG variables (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following ECG information will be collected:
  * Interpretation of the ECG (Normal/Abnormal/Borderline)
  * Heart rhythm
  * Presence of extrasystoles
  * Presence of conduction abnormalities
  * Evidence of left ventricular hypertrophy (LVH)
Sural nerve and tibial nerve amplitude (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  Sural nerve and tibial nerve amplitude will be measured in overall and in patients initiating a treatment with eplontersen
Biomarker results (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following biomarker results will be collected:
  * Serum TTR levels
  * Complete blood count
  * Hemoglobin
  * Troponin I
  * Cystatin
  * Creatinine
  * Reported glomerular filtration rate (GFR)
  * Albumin
  * Liver enzymes: alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), total bilirubin
  * N-terminal pro B-type natriuretic peptide (NT-proBNP)
  * Vitamin A level
  * Neurofilament light chain (NfL)
  * International normalized ratio (INR) test
Urine test results (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following test results will be collected:
  * Urine albumin-creatinine ratio (UACR)
  * Urine protein creatinine ratio (UPCR)
Clinical manifestations (signs and symptoms) of ATTR amyloidosis (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following clinical manifestations will be assessed:
  ischemic heart disease, acute myocardial infarction, heart failure, atrial fibrillation, arrhythmias, conduction system disease, aortic valve stenosis polyneuropathy, carpal tunnel syndrome, autonomic neuropathy, nephrotic syndrome, subnephrotic proteinuria, gastrointestinal dysfunction, chronic kidney disease / acute kidney injury, spinal stenosis, spinal stenosis surgery, hepatomegaly, ascites, oedema, other amyloidosis related manifestations (e.g., Popeye's sign, tendon rupture)
36-Item Short Form Health Survey Version 2 (SF-36v2) Physical Component Summary score (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  The SF-36v2 is a 36-item, generic health survey that provides scores for eight health domains (physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health) and two summary scores; the physical component summary (PCS) score and the mental component summary (MCS) score. Higher scores indicate a better health state.
Norfolk Quality of Life-Diabetic Neuropathy total score (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  The Norfolk QOL-DN is a 35-item, disease-specific instrument that provides scores for five domains (symptoms, large fiber neuropathy, small fiber neuropathy, autonomic neuropathy, and activities of daily living) and a total score. Higher scores indicate a worse health state.
Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  The KCCQ is a 23-item, disease-specific questionnaire that assesses seven domains (physical limitations, symptom stability, symptom frequency, symptom burden, self-efficacy, quality of life, and social limitation) and provides three summary scores (total symptom score, clinical summary score, and overall summary score). Higher scores indicate a better health state.
New York Heart Association (NYHA) classification (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  I=No symptoms; II=Symptoms with ordinary physical activity; III=Symptoms with less than ordinary physical activity; IV=Symptoms at rest.
National Amyloidosis Centre (NAC) ATTR staging or Mayo staging (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  For NAC staging, Stage I: N-terminal pro-brain natriuretic peptide (NT-proBNP) ≤3000 ng/L and estimated glomerular filtration rate (eGFR) ≥45 ml/min; Stage III: NT-proBNP >3000 ng/L and eGFR <45 ml/min; Stage IV:NT-proBNP ≥10,000 ng/L; Stage II: remainder of patients
  For Mayo staging, Stage I: Both and biomarker values are below the established thresholds; Stage II: Either troponin T or NT-proBNP is above the threshold; Stage III: Both troponin T and NT-proBNP biomarker values are above the threshold.
  Biomarker Thresholds: Troponin T: >0.05 mg/mL and NT-proBNP: >3000 pg/mL.
Familial amyloid polyneuropathy (FAP) (Coutinho) staging (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  Stage 0: No symptoms; Stage I: Unimpaired ambulation; mostly mild sensory, motor and autonomic neuropathy in the lower limbs; Stage II: Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk; Stage III: Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs.
Polyneuropathy disability (PND) score (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  Stage 0=No symptoms; Stage I=Sensory disturbances but preserved walking capabilities; Stage II=Impaired walking capacity, but ability to walk without a stick or crutches; Stage IIIA=Walking with help of 1 stick or crutch; Stage IIIB=Walking with the help of 2 sticks or crutches; Stage IV=confined to wheel chair or bedridden.
Left Ventricular Ejection Fraction (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  Left Ventricular Ejection Fraction will be measured in overall and in patients initiating a treatment with eplontersen
6-minute walk test (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  To address this objective, the distance walked in 6 minutes will be measured.
Charlson comorbidity index (CCI) and CCI components (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address CCI, most recent score and all CCI componenet will be measured
  * Myocardial infarction
  * Congestive heart failure
  * Peripheral vascular disease
  * Cerebrovascular disease
  * Dementia
  * Chronic pulmonary disease
  * Rheumatic disease
  * Peptic ulcer disease
  * Diabetes (None, Without chronic complications, With chronic complications)
  * Hemiplegia or paraplegia
  * Renal disease
  * Any malignancy, including lymphoma and leukemia, except malignant neoplasm of skin (None, Localized, Metastatic)
  * Liver disease (None, Mild, Moderate, Severe)
  * Metastatic solid tumor
  * Acquired immune deficiency syndrome (AIDS) / Human immunodeficiency virus (HIV)
Other comorbidities of interest (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following information will be collected:
  * Percentage of patients with depression
  * Percentage of patients with fibromyalgia
  * Percentage of patients with paraproteinemia
Healthcare resource utilization (overall and in patients initiating a treatment with eplontersen) | From time of enrollment for up to 7 years
  In order to address this objective, the following information will be collected:
  * Number of emergency department visits
  * Number of outpatient visits
  * Inpatient care/hospitalization general ward (non-intensive): number of inpatient stays, number of bed days
  * Inpatient care/hospitalization intensive ward: number of inpatient stays, number of bed days
Mortality (overall and in patients initiating a treatment with eplontersen) | Throughout study follow-up (up to 7 years)
  Mortality during study follow-up (all-cause, related to ATTR amyloidosis), overall and by NYHA/NAC or Mayo/FAP stage
Liver Disease and Live Transplant | From time of Enrollment for up to 7 Years
  * Liver disease (for patients with mild, moderate or severe liver disease: Child Pugh score, Child Pugh class, ascites, encephalopathy)
  * Liver transplantation (reason for transplant, type of transplant)

SECONDARY OUTCOMES:
Comparison of demographic and clinical characteristics of patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Demographics
  * mBMI
  * Medical history
  * Family history of ATTR amyloidosis
  * Time period between the first symptoms to date of diagnosis of ATTR amyloidosis
  * Time since diagnosis of ATTR amyloidosis
Comparison of findings from biopsy in patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Type of biopsy
  * Amyloid identification result (Positive, Negative, Inconclusive for amyloid)
  * Method of amyloid typing
  * Result of the biopsy (Normal/Abnormal)
  * Reason for considering the biopsy result abnormal
Comparison of findings from Cardiovascular magnetic resonance imaging (CMR) in patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments: extracellular volume (ECV), contrast use, left ventricular (LV) end-diastolic volume, LV end-systolic volume, LV ejection fraction, LV Mass Index, interventricular wall thickness, right ventricular Free Wall Thickness, LV Free Wall Thickness, left Atrial Volume Index, native T1 mapping, CMR result (Normal/Abnormal), reason for considering the result abnormal.
Comparison of findings from Echocardiography in patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments: LV ejection fraction, LV End Diastolic Volume, LV End Systolic Volume LV End Diastolic Dimension, LV End Systolic Dimension, Interventricular Septal, Thickness Diastole, Posterial Wall Thickness Diastole, Left Ventricular Mass Index, Left Atrial Volume, Left Atrial Volume Index, Mitral valve regurgitation, Aortic valve regurgitation, Tricuspid valve regurgitation, Pulmonic valve regurgitation, LV Outflow Gradient, Stroke Volume, Lateral early diastolic myocardial velocity (e' lateral), Medial early diastolic myocardial velocity (e' medial), Mitral E/e' Ratio, Early diastolic mitral inflow velocity (E), Late diastolic mitral inflow velocity (A), Mitral Peak E/A Ratio, Global LV longitudinal strain, Pulmonary artery systolic pressure, RV Free Wall Thickness Severity of Aortic stenosis, Severity of Mitral stenosis.
Comparison of ECG variables of patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Interpretation of the ECG (Normal/Abnormal/Borderline)
  * Heart rhythm
  * Presence of extrasystoles
  * Presence of conduction abnormalities
  * Evidence of left ventricular hypertrophy (LVH)
Comparison of findings from Bone tracer cardiac scintigraphyin patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments: Type of tracer, Heart to contralateral lung ratio (H/CL), Perugini grade, scintigraphy result (Normal/Abnormal), reason for considering the result abnormal.
Comparison of sural nerve and tibial nerve amplitude in patients prescribed eplontersen at any time during the observation eriod to patients on other ATTR treatments | Up to 7 years
  Sural nerve and tibial nerve amplitude will be compared in patients prescribed eplontersen at any time during the observation period to patients on other ATTR treatments
Comparison of biomarker results in patients prescribed eplontersen at any time during the observation eriod to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Serum TTR levels
  * Complete blood count
  * Hemoglobin
  * Troponin I
  * Cystatin
  * Creatinine
  * Reported glomerular filtration rate (GFR)
  * Albumin
  * Liver enzymes: alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), total bilirubin
  * N-terminal pro B-type natriuretic peptide (NT-proBNP)
  * Vitamin A level
  * Neurofilament light chain (NfL)
  * International normalized ratio (INR) test
Comparison of urine test results in patients prescribed eplontersen at any time during the observation eriod to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Urine albumin-creatinine ratio (UACR)
  * Urine protein creatinine ratio (UPCR)
Comparison of Clinical manifestations (signs and symptoms) of ATTR amyloidosis in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments: ischemic heart disease, acute myocardial infarction, heart failure, atrial fibrillation, arrhythmias, conduction system disease, aortic valve stenosis polyneuropathy, carpal tunnel syndrome, autonomic neuropathy, nephrotic syndrome, subnephrotic proteinuria, gastrointestinal dysfunction, chronic kidney disease / acute kidney injury, spinal stenosis, spinal stenosis surgery, hepatomegaly, ascites, oedema, other amyloidosis related manifestations (e.g., Popeye's sign, tendon rupture)
Comparison of 36-Item Short Form Health Survey Version 2 (SF-36v2) Physical Component Summary score in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  SF-36v2, physical component summary scores will be compared between patients treated with eplontersen and patients on other ATTR treatments.
Comparison of Norfolk Quality of Life-Diabetic Neuropathy total score in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  Norfolk Quality of Life-Diabetic Neuropathy total scores will be compared between patients treated with eplontersen and patients on other ATTR treatments.
Comparison of Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  Kansas City Cardiomyopathy Questionnaire (KCCQ) overall summary score will be compared in patients prescribed eplontersen to patients on other ATTR treatments
Comparison of New York Heart Association (NYHA) classification in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  New York Heart Association (NYHA) classification will be compared in patients prescribed eplontersen to patients on other ATTR treatments
Comparison of Familial amyloid polyneuropathy (FAP) (Coutinho) staging in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  FAP staging:
  Stage 0: No symptoms; Stage I: Unimpaired ambulation; mostly mild sensory, motor and autonomic neuropathy in the lower limbs; Stage II: Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk; Stage III: Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs.
Comparison of Left Ventricular Ejection Fraction in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  Left Ventricular Ejection Fraction will be compared in patients prescribed eplontersen to patients on other ATTR treatments
Comparison of Charlson comorbidity index (CCI) and CCI components in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  Charlson comorbidity index (CCI) and CCI components will be compared in patients prescribed eplontersen to patients on other ATTR treatments
Comparison of other comorbidities of interest in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Percentage of patients with depression
  * Percentage of patients with fibromyalgia
  * Percentage of patients with paraproteinemia
Comparison of healthcare resource utilization in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  The following outcomes will be compared between patients treated with eplontersen and patients on other ATTR treatments:
  * Number of emergency department visits
  * Number of outpatient visits
  * Inpatient care/hospitalization general ward (non-intensive): number of inpatient stays, number of bed days
  * Inpatient care/hospitalization intensive ward: number of inpatient stays, number of bed days
Comparison of mortality in patients prescribed eplontersen to patients on other ATTR treatments | Up to 7 years
  Mortality will be compared in patients prescribed eplontersen to patients on other ATTR treatments

OTHER OUTCOMES:
Risk factors for worsening ATTR progression | up to 7 years
  Factors associated with changes in clinical manifestations of ATTR amyloidosis, NYHA classification, NAC ATTR staging or Mayo staging, FAP (Coutinho) staging, PND score, LVEF, CCI and CCI components, and other comorbidities of interest will be identified.
Healthcare costs in patients with ATTR amyloidosis | Up to 7 years
  Average annual costs will be calculated based on available data in the different countries.
Serious adverse events in patients treated with ATTR amyloidosis treatments | Up to 7 years
  Serious adverse events in patients treated with ATTR amyloidosis treatments will be measured

CONTACTS AND LOCATIONS:
Locations (42):
- United States (24):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, New Brunswick, New Jersey
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Danville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Rimouski, Quebec
- Germany (8):
  - Research Site, Würzburg, Bavaria
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Hanover, Lower Saxony
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, Mainz, Rhineland-Palatinate
  - Research Site, Homburg, Saarland
  - Research Site, Berlin
- Spain (2):
  - Research Site, Bilbao, Basque Country
  - Research Site, Salamanca, Castille and León
- United Kingdom (3):
  - Research Site, Birmingham, West Midlands
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Plan to share only the redacted CSR synopsis
Supporting Information: CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Gillmore JD, Hahn K, Smith JG, Conceicao I, Tian Z, Grogan M, Pao C, Wittbrodt E, Jarbrink K, Papas MA, Davis MK. Rationale and Design of ANTHOLOGY: An ATTR Amyloidosis Real-World Evidence Program Aiming to Address Gaps in Amyloidosis Care. Cardiol Ther. 2025 Sep;14(3):477-490. doi: 10.1007/s40119-025-00402-y. Epub 2025 Mar 19. PMID 40108078